CLINICAL TRIAL: NCT03271359
Title: EMDR vs. PC For Motor Vehicle Accident Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trauma Institute & Child Trauma Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-GRE-3
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Trauma, Psychological; Motor Vehicle Accident
MeSH Terms: conditions — Psychological Trauma | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Eye movement desensitization and reprocessing (EMDR) arm (Experimental)
  Interventions: Behavioral: EMDR
- Progressive counting (PC) arm (Experimental)
  Interventions: Behavioral: PC

INTERVENTIONS:
Behavioral: EMDR — Initial EMDR session of up to three hours; about one week later, follow-up session of up to one hour
  Arms: Eye movement desensitization and reprocessing (EMDR) arm
Behavioral: PC — Initial PC session of up to three hours; about one week later, follow-up session of up to one hour
  Arms: Progressive counting (PC) arm

SUMMARY:
This is a randomized clinical trial comparing eye movement desensitization and reprocessing (EMDR) to progressive counting (PC) for volunteers from the community who are distressed by the memory of a motor vehicle accident. Participants will be assigned to the geographically nearest therapist, and then randomized to treatment condition.

ELIGIBILITY:
Inclusion Criteria:

* adult reporting distress related to motor vehicle accident-related trauma
* English-speaking

Exclusion Criteria:

* already in therapy in which the memory of interest is being actively addressed with a structured/focused trauma resolution method
* any obvious/urgent need for more comprehensive psychotherapy (based on initial screening interview)
* any indication of instability during interactions prior to the therapy session
* an average score on the Dissociative Experiences Scale of 30 or greater, if (as per follow-up questions) indicating a likely dissociative disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01-05 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in SUDS following treatment | Administered pre-treatment, two weeks post-treatment, and 12 weeks post-treatment
  Subjective Units of Distress Scale
Change in PRS following treatment | Administered pre-treatment, two weeks post-treatment, and 12 weeks post-treatment
  Problem Rating Scale
Change in PDS following treatment | Administered pre-treatment, two weeks post-treatment, and 12 weeks post-treatment
  PTSD Diagnostic Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Greenwald, Principal Investigator — Trauma Institute & Child Trauma Institute
Locations (1):
- Trauma Institute & Child Trauma Institute, Northampton, Massachusetts, United States